CLINICAL TRIAL: NCT00332878
Title: RCT of Stepping Stones Behavioural Intervention for HIV
Brief Title: Stepping Stones Program for Preventing HIV Infection in Residents of Rural South African Communities
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical Research Council, South Africa (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Tasnim Mohsam, Administrator, Medical Research Council, South Africa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01MH064882 (NIH); R01MH064882 (NIH); DAHBR 9A-ASI
Record Dates: First submitted 2006-06-01; First posted 2006-06-02 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: HIV Infections
Keywords: Behavioral Intervention; HIV; HSV2
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Stepping Stones
  Interventions: Behavioral: Stepping Stones
- 2 (Active Comparator): A 3 hour intervention on HIV and safer sex
  Interventions: Behavioral: stepping Stones short

INTERVENTIONS:
Behavioral: Stepping Stones — a comprehensive sexual and reproductive health promotion programme lasting about 50 hours comprising 13 content sessions of about 3 hours duration and 4 meetings of peer groups
  Arms: 1
Behavioral: stepping Stones short — 3 hour intervention on HIV and safer sex
  Arms: 2

SUMMARY:
This study will evaluate the effectiveness of Stepping Stones, an HIV-prevention education program, versus a brief HIV-focused intervention, in improving sexual health and preventing HIV infection in young residents of rural South African communities.

DETAILED DESCRIPTION:
HIV is arguably the most important problem currently facing the South African population. It is possible that biotechnology will eventually be able to lessen the disease's threat by introducing a vaccine or vaginal microbicide, but these are not expected to be available within the next 5 to 10 years. It is therefore extremely important to prevent HIV infection by modifying sexual behaviors. Voluntary counseling and testing have been shown to have an important impact on sexual behavior, but it is essential that other approaches to HIV prevention are developed and evaluated. Little research, however, has been done on behavioral interventions, relative to the amount of research that has been devoted to biotechnology development. Stepping Stones is an approach to HIV prevention that aims to improve sexual health through building stronger, more gender-equitable relationships with better communication between partners. This study will evaluate the effectiveness of the Stepping Stones program versus a brief HIV-focused intervention in improving sexual health and preventing HIV infection in young residents of rural South African communities.

Participants in this open-label study will be randomly assigned to take part in either the Stepping Stones program or the brief HIV-focused intervention (control). All participants will first attend a baseline study visit, which will include an interview and HIV testing. The control intervention will entail a single 2- to 3-hour meeting among same-sex peer groups, and will include exercises about HIV and safer sex practices that will be drawn from the Stepping Stones program. Stepping Stones will entail 17 sessions with same-sex peer groups, and will be implemented over a period of 3 to 12 weeks. Sessions will involve discussions on a variety of sexual health issues, including the following topics: reflections on love; sexual health joys and problems; body mapping; menstruation; contraception and conception, including infertility; sexual problems; unwanted pregnancy; HIV; STDs; safer sex; gender-based violence; motivations for sexual behavior; and dealing with grief and loss. Peer groups will come together for 3 of the 17 meetings to build assertive communication skills by leading presentations on exercises from the Stepping Stones program. HIV testing will be performed again after 12 and 24 months to assess program effectiveness. Face-to-face interviews will be held at Months 6, 12, and 24 to assess the impact of the intervention on behavior, attitude, and beliefs.

ELIGIBILITY:
Inclusion Criteria:

* Resident of the village in which individual is studying (i.e., not a migrant scholar)
* Mature enough to understand the study and the consent process

Exclusion Criteria:

* N/A

Ages: 16 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2801 (Actual)
Dates: Start 2003-03; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
HIV sero-incidence | 24 months post-baseline

SECONDARY OUTCOMES:
HSV-2 sero-incidence | 24 months post-baseline
correct condom use at last sex, number of partners, transactional sex, intimate partner violence, any casual partner, | 12 months and 24 months post-baseline

CONTACTS AND LOCATIONS:
Overall Officials: Rachel K. Jewkes, MBBS MSc MD, Principal Investigator — Medical Research Council, South Africa
Locations (1):
- Various villages in South Africa, Mthatha, Eastern Cape, South Africa

REFERENCES:
- [Background] Jewkes R, Nduna M, Levin J, Jama N, Dunkle K, Khuzwayo N, Koss M, Puren A, Wood K, Duvvury N. A cluster randomized-controlled trial to determine the effectiveness of Stepping Stones in preventing HIV infections and promoting safer sexual behaviour amongst youth in the rural Eastern Cape, South Africa: trial design, methods and baseline findings. Trop Med Int Health. 2006 Jan;11(1):3-16. doi: 10.1111/j.1365-3156.2005.01530.x. PMID 16398750
- [Derived] Jewkes R, Nduna M, Levin J, Jama N, Dunkle K, Puren A, Duvvury N. Impact of stepping stones on incidence of HIV and HSV-2 and sexual behaviour in rural South Africa: cluster randomised controlled trial. BMJ. 2008 Aug 7;337:a506. doi: 10.1136/bmj.a506. PMID 18687720